CLINICAL TRIAL: NCT05829369
Title: The Effects of Intrinsic Foot Muscle Strengthening Interventions on Balance, Proprioception, Foot Structure, and Fall Risk in Adults Over Age 65
Brief Title: Intrinsic Foot Muscle Strengthening Interventions for Older Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Springfield College (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: U01CE003495 (NIH)
Record Dates: First submitted 2023-01-31; First posted 2023-04-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Accidental Fall
Keywords: older adults; falls; feet; balance; proprioception; muscle strength

STUDY DESIGN:
Intervention Model Description: Randomized control trial with an effectiveness-implementation hybrid design Type I
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants are unable to be blinded to treatment they are receiving, but they will not be told interventions of other groups.
  Investigators who perform measurements are blinded to intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intrinsic foot muscle exercise (Experimental): This group will perform intrinsic foot muscle strengthening exercises
  Interventions: Other: Intrinsic foot muscle strengthening exercises
- Minimal Footwear (Active Comparator): This group will perform prescribed walking in and daily wear of minimally cushioned footwear
  Interventions: Other: Minimal footwear with prescribed walking
- Control (Sham Comparator): This group will be given a falls prevention brochure and seated upper extremity and lower extremity active range of motion activities.
  Interventions: Other: Control

INTERVENTIONS:
Other: Intrinsic foot muscle strengthening exercises — participants will perform specific toe and foot motions that recruit plantar intrinsic foot muscles, 3 sets of 10 for each exercise, 5 days per week
  Arms: Intrinsic foot muscle exercise
Other: Minimal footwear with prescribed walking — Participants will be provided minimal footwear. They will walk 30 minutes per day, 5 days per week, and be prescribed a gradual increased time in minimal footwear during daily activities (up to a maximum of 7.5 hours per day).
  Arms: Minimal Footwear
Other: Control — Participants will perform seated upper and lower extremity active range of motion activities 5 days per week. They will also be given a brochure on fall prevention tips.
  Arms: Control

SUMMARY:
Falls are the leading cause of injury in adults over age 65. Muscle weakness in the foot can lead to foot and toe deformities such as collapsed arches or bunions, which have been found to contribute to falls in adults over age 65. The current research study aims to investigate the effectiveness of two simple and affordable foot strengthening methods that may make a major impact on balance and fall prevention in older adults.

DETAILED DESCRIPTION:
Background: Falls are the leading cause of injury in adults 65 years and older. While causes of falls are multifactorial, foot function plays a vital role. The intrinsic foot muscles (IFM), those that originate and insert within the foot, provide stability and sensory input important for balance. Weakness or disuse of the IFM in older adults can contribute to faulty foot and toe alignment, which have been cited as independent predictors of falls. Wearing minimally cushioned footwear or performing strengthening exercises that target the IFM may improve these muscles' strength, endurance, proprioceptive qualities, and foot/toe structure, which may improve functional mobility and balance in older adults, and thus, prevent falls.

Purpose: The purpose of the proposed research is to analyze the effects of two IFM strengthening interventions (minimal footwear use or strengthening exercises) on IFM strength, proprioception, foot/toe structure, balance and functional mobility, and fall risk in older adults.

Design: Randomized control trial with an effectiveness-implementation hybrid design Type I

Methods: Adults ages > 65 years who can ambulate household distances with or without an assistive device who are determined to be at risk for falls will be invited to participate. Individuals with poor foot sensation, vestibular disorders, lower extremity amputation, injury or surgery to the lower extremities or lumbar spine in the previous 6 months, impaired cognitive ability to follow verbal and written instructions, and those who have participated in a fall prevention program in the past 6 months will be excluded. Following informed consent and initial screening, participants will be randomly allocated to one of three intervention groups (n=90, 30/group):

1. intrinsic foot muscle strengthening exercises
2. minimal footwear prescribed walking
3. control (will receive a fall prevention brochure and seated active motion exercises)

Participants will be encouraged to perform interventions 5 days/week for 16 weeks. After an initial in-person instruction session, participants will have 1 follow-up meeting to review instructions, after which they will receive bimonthly phone calls as a reminder to adhere to the intervention and to record any falls and related details. Participants will be asked to record intervention performance, daily step count (measured by pedometer), and falls in provided diaries. Balance, functional mobility, and fall risk will be measured using the Mini-BesTest, proprioception will be measured using the Lower Extremity Position Test, foot and toe structure will be measured using navicular drop and valgus angle of the 1st metatarsophalangeal joint. Cross sectional area (cm2) of the abductor hallucis, flexor hallucis brevis, flexor digitorum brevis, and quadratus plantae muscles will be measured using ultrasound imaging. Measures regarding balance and functional mobility, proprioception, foot/toe structure, and muscle cross sectional area will occur at baseline, 8 and 16 weeks, and 1 year. Following the 16-week intervention period, participants will be encouraged to continue their intervention twice per week. Ongoing falls diaries and bimonthly phone calls from researchers will occur for 12 months after baseline to record long-term fall rate (falls per person per year). In addition, a process evaluation will be performed regarding participant impressions of the interventions and other study activities to inform future research and clinical implementation.

Data Analysis: a 4 group x 4 time point repeated measures analysis of covariance (ANCOVA) will be used to assess changes in balance, and functional mobility, proprioception, foot/toe structure, and muscle cross sectional area. Falls data will be measured as the rate of falls per person in a 12-month period beginning with the date of the baseline measure, and change in fall risk status will be assessed using Mini-BesTest scores. Implementation data will undergo both quantitative and qualitative analyses.

Significance: Intrinsic foot muscle strengthening interventions have seldom been studied in older adults and their effects and mechanism are not established. This will be the first study to assess the effects of these interventions on proprioception in older adults, the first to use ultrasound imaging measurement following intrinsic foot muscle strengthening in older adults, and the first study to analyze the long-term effects on falls after the performance of these specific interventions. The interventions assessed in this research proposal are simple, safe, and affordable and may have a major impact on functional mobility and reduction of falls for older adults.

ELIGIBILITY:
Inclusion Criteria:

* Can ambulate household distances (16 meters) with or without an assistive device
* Have fall risk based on a "yes" to any of the Three Key Questions Do you feel unsteady when standing or walking? Do you worry about falling? Have you fallen in the past year? OR
* Have a fall risk based on Timed Up and Go score (> 12 seconds)

Exclusion Criteria:

* poor foot sensation (Semmes-Weinstein)
* lower extremity amputations
* lumbar spine or lower extremity injury or surgery in the past 6 months
* impaired cognitive ability to follow verbal or written instructions (MMSE)
* vestibular disorders
* based on self-report and/or the Vestibular Screening Tool (score > 4)
* participation in a fall prevention program in the previous 6 months

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-12-16 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in Mini BesTest scores | Baseline
  a comprehensive measure of balance, gait, and functional mobility (max score 28 and indicates good balance/mobility and low fall risk)
Change in Mini BesTest scores | 8 weeks post intervention
  a comprehensive measure of balance, gait, and functional mobility (max score 28 and indicates good balance/mobility and low fall risk)
Change in Mini BesTest scores | 16 weeks post intervention
  a comprehensive measure of balance, gait, and functional mobility (max score 28 and indicates good balance/mobility and low fall risk)
Change in Mini BesTest scores | 1 year post intervention
  a comprehensive measure of balance, gait, and functional mobility (max score 28 and indicates good balance/mobility and low fall risk)
Change in intrinsic foot muscle cross-sectional area/strength | Baseline
  real-time ultrasound imaging will measure muscle size (cross-sectional area) of the abductor hallucis, flexor hallucis brevis, flexor digitorum brevis, quadratus plantae, and abductor digiti minimi muscles of the right foot
Change in intrinsic foot muscle cross-sectional area/strength | 8 weeks post intervention
  real-time ultrasound imaging will measure muscle size (cross-sectional area) of the abductor hallucis, flexor hallucis brevis, flexor digitorum brevis, quadratus plantae, and abductor digiti minimi muscles of the right foot
Change in intrinsic foot muscle cross-sectional area/strength | 16 weeks post intervention
  real-time ultrasound imaging will measure muscle size (cross-sectional area) of the abductor hallucis, flexor hallucis brevis, flexor digitorum brevis, quadratus plantae, and abductor digiti minimi muscles of the right foot
Change in intrinsic foot muscle cross-sectional area/strength | 1 year post intervention
  real-time ultrasound imaging will measure muscle size (cross-sectional area) of the abductor hallucis, flexor hallucis brevis, flexor digitorum brevis, quadratus plantae, and abductor digiti minimi muscles of the right foot

SECONDARY OUTCOMES:
Change in hallux valgus angle | Baseline
  a goniometer will be used to measure the angle of the 1st metatarsophalangeal joint of the right foot
Change in hallux valgus angle | 8 weeks post intervention
  a goniometer will be used to measure the angle of the 1st metatarsophalangeal joint of the right foot
Change in hallux valgus angle | 16 weeks post intervention
  a goniometer will be used to measure the angle of the 1st metatarsophalangeal joint of the right foot
Change in hallux valgus angle | 1 year post intervention
  a goniometer will be used to measure the angle of the 1st metatarsophalangeal joint of the right foot
Change in navicular drop measure | Baseline
  the Navicular Drop Test will measure the amount of foot pronation in sitting and standing
Change in navicular drop measure | 8 weeks post intervention
  the Navicular Drop Test will measure the amount of foot pronation in sitting and standing
Change in navicular drop measure | 16 weeks post intervention
  the Navicular Drop Test will measure the amount of foot pronation in sitting and standing
Change in navicular drop measure | 1 year post intervention
  the Navicular Drop Test will measure the amount of foot pronation in sitting and standing
Change in proprioception measure | Baseline
  The Lower Extremity Proprioception Test will be used to capture proprioception of the foot, ankle, and knee in sitting
Change in proprioception measure | 8 weeks post intervetion
  The Lower Extremity Proprioception Test will be used to capture proprioception of the foot, ankle, and knee in sitting
Change in proprioception measure | 16 weeks post intervention
  The Lower Extremity Proprioception Test will be used to capture proprioception of the foot, ankle, and knee in sitting
Change in proprioception measure | 1 year post intervention
  The Lower Extremity Proprioception Test will be used to capture proprioception of the foot, ankle, and knee in sitting

CONTACTS AND LOCATIONS:
Overall Officials: Erin Futrell, PhD, Principal Investigator — Springfield College
Locations (1):
- Springfield College, Springfield, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided